CLINICAL TRIAL: NCT01096407
Title: The Role of COX-2 Mediated Prostaglandin Production on Paclitaxel-Induced Myalgias and Arthralgias.
Brief Title: Role of Biomarkers in Muscle Pain and Joint Pain in Patients With Solid Tumors Receiving Paclitaxel
Status: Terminated | Type: Observational
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jill Gilbert, MD, Associate Professor of Medicine; Director, Hematology/Oncology Fellowship Program; Section Chief, Solid Tumor Oncology; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC SUPP 0928; P30CA068485 (NIH); VU-VICC-SUPP-0928
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Arthralgia; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: pain; arthralgia; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Arthralgia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Paclitaxel-Induced Myalgias/Arthralgias
  Interventions: Other: laboratory biomarker analysis; Other: questionnaire administration; Procedure: assessment of therapy complications

INTERVENTIONS:
Other: laboratory biomarker analysis — Collection of urine samples
Other: questionnaire administration — Completion of questionnaires
Procedure: assessment of therapy complications — An assessment will be completed.

SUMMARY:
RATIONALE: Learning about pain in patients with cancer receiving paclitaxel may help plan treatment and may help patients live more comfortably. Studying samples of urine from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to muscle and joint pain.

PURPOSE: This phase I trial is studying the role of biomarkers in muscle pain and joint pain in patients with solid tumors receiving paclitaxel.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the change in urinary prostaglandin E metabolite (PGE-M) level after paclitaxel treatment in patients with a variety of solid tumor malignancies.
* To determine whether a change in PGE-M level correlates with paclitaxel dose.
* To determine whether the change in urinary PGE-M level correlates with patient reporting of pain, as measured by a visual analog scale and the Brief Pain Inventory short form (BPI-SF).

Secondary

* To determine whether leukotriene levels are affected by paclitaxel treatment.

OUTLINE: At baseline (prior to the first dose of paclitaxel), patients complete a questionnaire about their baseline pain symptoms (including the Brief Pain Inventory short form and the visual analog scale); cigarette smoking status and second-hand smoke exposure; and routine use of any pain medications (including NSAIDs, selective COX-2 inhibitors, and opioid analgesics), corticosteroids, or leukotriene antagonists (montelukast or zafirlukast). Patients also complete questionnaires about their pain daily on days 2-7 after paclitaxel administration.

Urine samples are collected at baseline for urinary prostaglandin E metabolite (PGE-M), urinary leukotriene E_4 (LTE_4), and urinary cotinine levels and on day 4 for urinary PGE-M and LTE_4 levels.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Solid malignancy of any type
* Patients must be scheduled to receive their first dose of paclitaxel at Vanderbilt-Ingram Cancer Center

  * Any paclitaxel-containing regimen or dosing schedule is allowed

PATIENT CHARACTERISTICS:

* Not pregnant
* Accessible for follow-up
* Able to submit urine samples
* Able to complete questionnaires

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients that will be treated with paclitaxel.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change in urinary PGE-M level after paclitaxel treatment | Day 1 before paclitaxel treatment and day 4, after treatment
  Change in amount of PGE-M in the urine from before administration of paclitaxel to 4 days after treatment.

SECONDARY OUTCOMES:
Correlation of change in urinary PEG-M level and paclitaxel dose | Day 1 before paclitaxel treatment and day 4, after treatment
  Inter-relationship between the dose of paclitaxel and the change in level of urinary PEG-M from before treatment compared to day 4 of paclitxel treatment
Correlation of urinary PEG-M level with pain | day 1 before paclitaxel treatment and day 4, after treatment
  Inter-relationship between the level of urinary PEG-M level with level of pain, measured from before treatment compared to day 4 after paclitaxel treatment. Pain is measured on the Brief Pain Inventory (BPI). The BPI consists of 7 questions about interference of pain in daily life, answered on a scale of 0 (does not interfere) to 10 (completely interferes). The summary score is the average of the 7 scores, with higher scores indicating greater interference with pain.
Change in urinary luekotriene E_4 level after paclitaxel treatment | day 1 before paclitaxel treatment and day 4, after treatment
  Inter-relationship be the level of urinary luekotriene E_4 from before treatment compared to day 4 after paclitaxel treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jill Gilbert, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee